CLINICAL TRIAL: NCT05261490
Title: A Phase Ⅰ/Ⅱ Study of TTI-622 in Combination With Pegylated Liposomal Doxorubicin in Patients With Platinum-Resistant Ovarian Cancer
Brief Title: Study of Maplirpacept (PF-07901801) in Combination With PLD in Patients With Platinum-Resistant Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A business decision was made by Pfizer to terminate and remove the Phase 2 expansion of this study for administrative reasons. The reason for study termination is not due to any safety concerns or requests from regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TTI-622-02; C4971002 (Other: Alias Study Number)
Record Dates: First submitted 2021-11-22; First posted 2022-03-02 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer; Ovarian Neoplasms; Ovarian Carcinoma; Fallopian Tube Cancer; Epithelial Ovarian Cancer; Primary Peritoneal Carcinoma
Keywords: Epithelial Ovarian Cancer (EOC); Ovarian Cancer; Platinum-Resistant Ovarian Cancer; Cluster of Differentiation 47 (CD47); maplirpacept (PF-07901801); TTI-622; Doxorubicin; Immune-oncology; chemotherapy; anti-SIRPα therapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — liposomal doxorubicin; 1-dodecylpyridoxal

STUDY DESIGN:
Intervention Model Description: Phase 1/2 (dose escalation and dose expansion)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental): In the Phase 1 (dose escalation):
  Cycle 1 for dose levels 1 and 2, maplirpacept (PF-07901801) will be administered on Day 1, Day 8, Day 15 and Day 22 in combination with PLD on Day 1 of 28-day cycle. Beginning with Cycle 2 at dose levels 1 and 2, maplirpacept (PF-07901801) will be administered on Day 1 and Day 15 in combination with PLD on Day 1 of 28-day cycles. For Phase 1, dose level 3, maplirpacept (PF-07901801) will be administered on Day 1 and Day 15 in combination with PLD on Day 1 of 28-day cycles. Dose level 3 will be biweekly regimen from the start.
  Interventions: Drug: maplirpacept (PF-07901801); Drug: Pegylated Liposomal Doxorubicin (PLD)
- Phase 2: Dose Expansion (Experimental): In the Phase 2 (dose expansion):
  maplirpacept (PF-07901801) will be administered with selected dose from the escalation phase by intravenous infusion on Days 1, 8, 15 and 22 in Cycle 1, and then on Days 1 and 15 in subsequent cycles in combination with Pegylated Liposomal Doxorubicin 40 mg/m2 by intravenous infusion on Day 1 of each 28-day cycle.
  Interventions: Drug: maplirpacept (PF-07901801); Drug: Pegylated Liposomal Doxorubicin (PLD)

INTERVENTIONS:
Drug: maplirpacept (PF-07901801) — PF-07901801 Escalation (3-dose-level 12, 24, and 48 mg/kg), in combination with Pegylated Liposomal Doxorubicin (40mg/m2) will be administered by intravenous infusion.
  Other Names: TTI-622
Drug: Pegylated Liposomal Doxorubicin (PLD) — RP2D of maplirpacept (PF-07901801) biweekly of maplirpacept (PF-07901801) from Phase 1 escalation in combination with pegylated liposomal doxorubicin 40mg/m2
  Other Names: PLD

SUMMARY:
Pegylated liposomal doxorubicin (PLD), a type of chemotherapy, is a standard treatment option for patients with platinum-resistant ovarian cancer. However, despite being consider a standard treatment option, the clinical benefit of chemotherapy alone for these patients is small. Historically, response rates for PLD monotherapy have only ranged from 12 to 35% with a high likelihood of recurrence within months after treatment initiation. Although bevacizumab (BEV), an anti-new-vascular growth monoclonal antibody has been approved by FDA to combine with standard chemotherapy (e.g., PLD) for platinum-resistant recurrent ovarian cancer, there are still many restrictions or contraindications preventing certain women from receiving bevacizumab's combination treatment. The goal of this study is to improve upon the activity of PLD in a safe manner to provide a more effective therapeutic option for this group of patients.

The purpose of this study is to assess maplirpacept (PF-07901801) administered in combination with PLD in patients with platinum-resistant ovarian cancer and for whom PLD is a reasonable treatment option. The first portion of the study will evaluate the safety of increasing dose levels of maplirpacept (PF-07901801) in combination with PLD at 40 mg/m2 in patients with platinum-resistant EOC (epithelial ovarian cancer). This is a group of cancer, including ovarian, peritoneal, and fallopian tube malignancy. The aim of the first portion of the study is to establish a combination regimen for further assessment in a dose expansion cohort.

The study will consist of a 28-day screening period to ensure participants are qualified for the study treatment plan. During the treatment period, patients will receive maplirpacept (PF-07901801) in combination with PLD in 28-day cycles until their disease progresses or unacceptable toxicity develops. There will be a long-term follow-up period in this study to assess overall survival (length of time since start of treatment patients are alive).

DETAILED DESCRIPTION:
Pegylated liposomal doxorubicin (PLD) is a standard treatment option for patients with platinum-resistant ovarian cancer who are not candidates for chemotherapy in combination with bevacizumab. However, despite being consider a standard treatment option, the clinical benefit of chemotherapy for this patient population is small. The goal of this clinical trial is to improve upon the activity of PLD in a safe manner to provide a more effective therapeutic option for this group of patients.

C4971002 (TTI-622-02) is a multi-center, open-label study designed to evaluate maplirpacept (PF-07901801) administered in combination with PLD in patients with platinum-resistant ovarian cancer and for whom PLD is a reasonable treatment option. The first portion of the study will evaluate the safety of increasing dose levels of maplirpacept (PF-07901801) in combination with PLD at 40 mg/m2 in patients with platinum-resistant EOC, including ovarian, peritoneal and fallopian tube malignancy, and establish a combination regimen for further evaluation in a dose expansion cohort. The study will consist of a 28-day screening period, a treatment period in which patients will receive maplirpacept (PF-07901801) in combination with PLD in 28-day cycles until documentation of objective disease progression or development of unacceptable toxicity, and a long-term follow-up period to assess overall survival.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Histologically-confirmed epithelial ovarian cancer (EOC), fallopian tube carcinoma (FTC) or primary peritoneal carcinomas (PPC).
* Platinum-resistant recurrent (disease progression ≤6 months after the most recent platinum-based treatment regimen (date calculated from the last administered dose of platinum) or the participant is no longer able to receive.

or declined treatment with platinum-based chemotherapy.

* Progression with standard of care therapies, including platinum-based therapies, poly ADP ribose polymerase (PARP) inhibitors or bevacizumab in the platinum-sensitive setting or intolerability to such therapies or patient refusal
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Adequate organ and hematologic function
* No more than four prior treatment regimens for platinum-resistant disease
* All adverse events from prior treatment must be the Common Terminology Criteria for Adverse Events (NCI CTCAE) v5 Grade ≤ 1, except alopecia and stable neuropathy, which must have resolved to Grade ≤ 2 or baseline.

Key Exclusion Criteria:

* Platinum-refractory disease (defined as progression on or within 3 months of completing primary first-line platinum-based treatment)
* Non-epithelial histology, including malignant mixed Mullerian tumors
* Ovarian tumors with low malignant potential (i.e., borderline tumors), low grade serous ovarian cancer or carcinosarcoma
* History of acute coronary syndromes.
* History of or current Class II, III, or IV heart failure.
* History or evidence of known central nervous system (CNS) metastases or carcinomatous meningitis.
* Significant bleeding disorders, vasculitis or a significant bleeding episode from the Gastrointestinal (GI) tract.
* History of severe hypersensitivity reactions to antibodies.
* Systemic steroid therapy.
* History or autoimmune disease that has required systemic treatment with disease-modifying agents, corticosteroids, or immunosuppressive drugs.
* Prior organ transplantation including allogenic or autologous stem cell transplantation
* Prior treatment with anti-cluster of differentiation 47 (CD47) or anti-SIRPα therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Baptist Hospital of Miami, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Orlando Health Cancer Institute Gynecologic Cancer Center, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Michigan Healthcare Professionals PC, Dearborn, Michigan
  - Michigan Healthcare Professionals PC, Farmington Hills, Michigan
  - Michigan Healthcare Professionals PC, Royal Oak, Michigan
  - Michigan Healthcare Professionals PC, Sterling Heights, Michigan
  - Cleveland Clinic taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio
  - Oklahoma Cancer Specialist and Research Institute. LLC, Tulsa, Oklahoma
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center-Investigational Drug Services, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - oncology Consultants, P.A., Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=TTI-622-02

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 phases of the study: Phase 1 and 2. Due to business decision the study was terminated, and Phase 2 was not conducted. Hence, results in all sections are reported only for Phase 1 of the study and not for Phase 2.
Pre-assignment Details: A total of 10 participants were enrolled and treated in the study (Phase 1).
Groups:
- Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + Pegylated Liposomal Doxorubicin (PLD): Participants received Maplirpacept 12 milligram per kilogram (mg/kg) by intravenous (IV) infusion on Days 1, 8, 15 and 22 of the 28-day for Cycle 1 and on Days 1 and 15 of subsequent 28-day cycles (Cycle 2 onward). Participants in combination received PLD 40 milligram per meter square (mg/m^2) intravenously on Day 1 of each 28-day cycle.
- Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD: Participants received Maplirpacept 24 mg/kg by IV infusion on Days 1, 8, 15 and 22 of the 28-day for Cycle 1 and on Days 1 and 15 of subsequent 28-day cycles (Cycle 2 onward). Participants in combination received PLD 40 mg/m^2 intravenously on Day 1 of each 28-day cycle.
- Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD: Participants received Maplirpacept 48 mg/kg by IV infusion on Days 1 and 15 of each 28-day cycle. Participants in combination received PLD 40 mg/m^2 intravenously on Day 1 of each 28-day cycle.
Period: Overall Study
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + Pegylated Liposomal Doxorubicin (PLD) | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Started | 3 | 3 | 4
Treated | 3 | 3 | 4
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 4
Not completed — Other | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 1 | 4
Not completed — Death | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who received at least one dose of Maplirpacept.
Groups:
- Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD: Participants received Maplirpacept 12 mg/kg by IV infusion on Days 1, 8, 15 and 22 of the 28-day for Cycle 1 and on Days 1 and 15 of subsequent 28-day cycles (Cycle 2 onward). Participants in combination received PLD 40 mg/m^2 IV on Day 1 of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (13.05) | 66.3 (3.79) | 67.3 (7.80) | 66.8 (7.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 10
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 4 | 7
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 2 | 3 | 3 | 8
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as hematologic and/or non-hematologic treatment-emergent adverse event (TEAE) that occurred during the 28-day Cycle 1 and were judged by the investigator as related to Maplirpacept or the combination of Maplirpacept and PLD. Adverse events (AEs) that were in the opinion of the investigator attributable exclusively to intravenous infusion of PLD or any PLD prophylaxis medication were not considered a DLT.
Time Frame: Cycle 1 (28 days)
Population: DLT evaluation population set included all participants in Phase 1 who either experienced DLT after at least one dose of Maplirpacept or did not experience a DLT and received the full dose of PLD and at least two infusions of Maplirpacept and completed safety evaluations during the 28-day Cycle 1 DLT period.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Participants | 0 | 0 | 0

2. Secondary Outcome: Phase 1: Number of Participants With TEAEs, Serious TEAEs, >=3 Grade TEAEs, Treatment Related TEAEs, Treatment Related Serious TEAEs and >=3 Grade Treatment Related TEAEs
Description: AE: untoward medical occurrence or the worsening of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to study treatment. TEAEs: event that occurred or worsened on or after start of Maplirpacept up to 30 days (+5) after last dose of study treatment or 1 day before starting day of new anti-cancer drug therapy; includes serious and all non-serious AEs. Serious AE: AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged in participant hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly. AEs' severity graded using common terminology criteria for AEs (CTCAE) v 5.0; grade 3= severe; grade 4= life-threatening; grade 5= death. Treatment-related AE: untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to drug was assessed by investigator.
Time Frame: From start of treatment up to 30 days (+5) after last dose of study treatment or 1 day before starting day of new anti-cancer drug therapy whichever occurred first (up to approximately 33 weeks; maximum exposure of study treatment = 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Participants
  TEAEs | 3 | 3 | 4
  Serious-TEAEs | 1 | 0 | 1
  Grade >= 3 TEAEs | 3 | 2 | 3
  Treatment-Related TEAEs, any study drug | 3 | 3 | 4
  Serious Treatment-Related TEAEs, any study drug | 0 | 0 | 1
  Grade >=3 Treatment-Related TEAEs, any study drug | 2 | 1 | 3

3. Secondary Outcome: Phase 1: Change From Baseline in Diastolic and Systolic Blood Pressure (BP) at End of Treatment
Description: BP was measured in millimeter of mercury (mmHg).
Time Frame: Baseline (prior to the start of study treatment on Day 1 Cycle 1), End of treatment (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
mmHg
  Diastolic BP | 7.3 (17.21) | -1.7 (8.08) | -12.5 (14.82)
  Systolic BP | 5.3 (22.23) | -11.0 (4.58) | -3.0 (8.76)

4. Secondary Outcome: Phase 1: Change From Baseline in Respiratory Rate at End of Treatment
Description: Respiratory rate was measured in breaths per minute (breaths/ min).
Time Frame: Baseline (prior to the start of study treatment on Day 1 Cycle 1), End of treatment (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Mean (Standard Deviation); unit: Breaths/ min
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Breaths/ min | 0.0 (0.00) | -1.3 (1.15) | 1.0 (1.15)

5. Secondary Outcome: Phase 1: Change From Baseline in Pulse Rate at End of Treatment
Description: Pulse rate was measured in beats per minute (beats/min).
Time Frame: Baseline (prior to the start of study treatment on Day 1 Cycle 1), End of treatment (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Mean (Standard Deviation); unit: Beats/ min
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Beats/ min | -4.3 (17.50) | -2.3 (15.31) | -8.0 (13.29)

6. Secondary Outcome: Phase 1: Change From Baseline in Temperature at End of Treatment
Description: Temperature was measured in degree Celsius (C).
Time Frame: Baseline (prior to the start of study treatment on Day 1 Cycle 1), End of treatment (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Mean (Standard Deviation); unit: Degree C
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Degree C | 0.3 (0.46) | -0.3 (0.25) | 0.1 (0.09)

7. Secondary Outcome: Phase 1: Change From Baseline in Weight at End of Treatment
Description: Weight was measured in kilogram (kg).
Time Frame: Baseline (prior to the start of study treatment on Day 1 Cycle 1), End of treatment (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
kg | -0.7 (1.74) | -4.6 (1.89) | -1.6 (4.90)

8. Secondary Outcome: Part 1: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Standard 12-lead ECGs utilizing limb leads were used to interpret normal and abnormal results, QT interval. ECG was performed after the participant had rested quietly for at least 10 minutes in a supine position. Clinical significance of ECG abnormalities were determined by the investigator.
Time Frame: During study treatment, (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Participants | 0 | 0 | 0

9. Secondary Outcome: Phase 1: Phase 1: Number of Participants With Shift to Grade 3/4 in Serum Chemistry Parameters Abnormalities From Baseline to Post-baseline During the Study Treatment
Description: Serum chemistry tests included determination of the following parameters: glucose, sodium, potassium, calcium, chloride, phosphate, bicarbonate, blood urea nitrogen or urea, creatinine, total protein, albumin, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, indirect bilirubin, uric acid, calcium, magnesium, and lactate dehydrogenase (LDH). The serum chemistry parameters were graded using CTCAE version 5.0. The intensity was assigned a grade of 1-5 using the following CTCAE guidelines: grade 1= mild; grade 2= moderate; grade 3= severe; grade 4= life-threatening; grade 5= death. In this outcome measure number of participants with at least 1 event of shift to grade 3 or 4 in serum chemistry parameters abnormalities from baseline to post-baseline during study treatment are reported.
Time Frame: Baseline to post-baseline during study treatment (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Participants | 0 | 0 | 0

10. Secondary Outcome: Phase 1: Number of Participants With Shift to Grade 3/4 in Hematology Parameters Abnormalities From Baseline to Post-baseline During the Study Treatment
Description: Hematology tests included determination of the following parameters: hemoglobin, hematocrit, platelets, white blood cells (WBC), neutrophils, lymphocytes, eosinophils, basophils, monocytes, WBC with automated 5-part differential, red blood cells (RBC), absolute reticulocytes, reticulocytes percentage (%), erythrocyte mean corpuscular hemoglobin (MCH), erythrocyte mean corpuscular volume (MCV), and red cell distribution width (RDW). Clinical significance was determined by the investigator. The hematology parameter was graded using CTCAE version 5.0. The intensity was assigned a grade of 1-5 using the following CTCAE guidelines: grade 1= mild; grade 2= moderate; grade 3= severe; grade 4= life-threatening; grade 5= death. In this outcome measure number of participants with at least 1 event of shift to grade 3 or 4 in hematology parameters abnormalities from baseline to post-baseline during study treatment are reported.
Time Frame: Baseline to post-baseline during study treatment (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Participants
  Neutrophil count decreased | 2 | 1 | 3
  White blood cell decreased | 2 | 0 | 2
  Lymphocyte count decreased | 1 | 0 | 2
  Platelet count decreased | 1 | 0 | 2

11. Secondary Outcome: Phase 1: Number of Participants With Dose Delay
Description: Dose delay was the difference between the actual time between two consecutive non-zero doses and the planned time between the same two consecutive non-zero doses. In this outcome measure number of participants with any event of dose delay are reported.
Time Frame: During study treatment, (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Participants | 2 | 0 | 3

12. Secondary Outcome: Phase 1: Number of Participants Who Discontinued Study Treatment Due to TEAE
Description: In this outcome measure number of participants who discontinued study treatment due to TEAE are reported. TEAEs: event that occurred or worsened on or after start of Maplirpacept up to 30 days (+5) after last dose of study treatment or 1 day before starting day of new anti-cancer drug therapy; includes serious and all non-serious AEs.
Time Frame: During study treatment, (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Participants | 2 | 0 | 1

13. Secondary Outcome: Phase 1: Progression Free Survival (PFS), Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1
Description: PFS: time from the first Maplirpacept infusion (Cycle 1 Day 1) to disease progression (PD) or death of any cause, whichever occurred first. Participants who completed or discontinued the study without PD or death, as well as participants who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date or last adequate assessment prior to the start date of alternate anti-cancer therapy. If date of progression occurred on the same date as the start of new anticancer therapy, the progression was counted as an event. PD per RECIST v1.1: at least a 20% increase in the sum of longest diameter (LD) of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of 1 or more new lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From first Maplirpacept infusion till PD or death or censoring date, whichever occurred earlier (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Months | 5.3 [1.6 to NA] — Upper limit of 95% confidence interval (CI) could not be estimated because of insufficient number of participants with events. | 1.7 [1.4 to NA] — Upper limit of 95% CI could not be estimated because of insufficient number of participants with events. | 3.8 [3.6 to NA] — Upper limit of 95% CI could not be estimated because of insufficient number of participants with events.

14. Secondary Outcome: Phase 1: Overall Survival (OS)
Description: OS was defined as the time from the first Maplirpacept infusion (Cycle 1 Day 1) to death of any cause. Participants without death date at the time of analysis were censored at their last known alive date. Analysis was planned to be performed using Kaplan-Meier method. However, the study was terminated prior to achieving meaningful number of events, hence Kaplan-Meier analysis was not conducted. In this outcome measure number of days from first Maplirpacept infusion until death for each participant (who had death as an event) is reported individually.
Time Frame: From first Maplirpacept infusion till death or censoring date, whichever occurred earlier (maximum up to 32 weeks)
Population: SAS included all participants who received at least one dose of Maplirpacept. "Number of Participants Analyzed" signifies participants with death as an event [0= no participant with event] and "Number Analyzed" signifies participants evaluable for specified rows. Since there were insufficient participants with event, data could not be summarized as planned by Kaplan-Meier analysis and have been reported for each participant who had event in applicable reporting arms.
Measure: Number; unit: Days
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 1 | 2 | 0
Days
  Participant 1: number analyzed (Participants) | 1 | 0 | 0
  Participant 1 | 138 |  |
  Participant 2: number analyzed (Participants) | 0 | 1 | 0
  Participant 2 |  | 150 |
  Participant 3: number analyzed (Participants) | 0 | 1 | 0
  Participant 3 |  | 204 |

15. Secondary Outcome: Phase 1: Phase 1: Disease Control Rate (DCR), Per RECIST v1.1
Description: DCR: percentage of participants who had achieved complete response (CR), partial response (PR), or stable disease (SD) lasting at least 12 weeks. According to RECIST v1.1 criteria: CR = disappearance of all target lesions, any pathological lymph nodes (whether target or on-target) must have reduction in short axis to <10 mm; PR = at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; SD = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started; PD = at least a 20% increase in the sum of LD of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions.
Time Frame: as for outcome 13
Population: SAS included all participants who received at least one dose of Maplirpacept.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 3 | 3 | 4
Percentage of participants | 66.7 [20.8 to 93.9] | 0.0 [0.0 to 56.1] | 50.0 [15.0 to 85.0]

16. Secondary Outcome: Phase 1: Duration of Response (DOR)
Description: DOR: for participants who achieved a confirmed CR or PR; defined as time from the date of first documented response (CR or PR) to the date of documented progression or death of any cause after achieving response. Participants who completed or discontinued the study without PD or death, as well as participants who received alternate anti-cancer therapy prior to PD, was censored at their last adequate response assessment date or last adequate assessment prior to start date of alternate anti-cancer therapy. CR=disappearance of all target lesions, any pathological lymph nodes must have reduction in short axis to <10 mm; PR=at least 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; PD= at least 20% increase in the sum of LD of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of 1 or more new lesions.
Time Frame: From time of first documented CR or PR to progression or death or censoring date, whichever occurred earlier (maximum up to 32 weeks
Population: Analysis of this outcome measure was to be evaluated in participants with confirmed CR or PR. Here, "Number of Participants Analyzed" = '0' signifies that no participant had confirmed CR or PR in any reporting arm. Hence, outcome measure not analyzed.
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of treatment up to 30 days (+5) after last dose of study treatment (up to approximately 33 weeks; maximum exposure of study treatment = 32 weeks)
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set included all participants who received at least one dose of Maplirpacept.
Arm/Group | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD (N=3) | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD (N=3) | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD (N=4)
Gait disturbance (General disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Maplirpacept (PF-07901801) 12 mg/kg + PLD (N=3) | Phase 1: Maplirpacept (PF-07901801) 24 mg/kg + PLD (N=3) | Phase 1: Maplirpacept (PF-07901801) 48 mg/kg + PLD (N=4)
Nausea (Gastrointestinal disorders) | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 1 | 3
Platelet count decreased (Investigations) | 2 | 1 | 3
Blood lactate dehydrogenase increased (Investigations) | 1 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 3
Gait disturbance (General disorders) | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 2
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Pyrexia (Investigations) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Candida infection (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vulval disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to business decision the study was terminated, and Phase 2 of the study was not conducted. Hence, none of the section reports results for Phase 2 of the study. Data reported is only for Phase 1 of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT05261490/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT05261490/SAP_001.pdf